CLINICAL TRIAL: NCT05074498
Title: A Seamless Phase 1b/2a Double-blind, Randomized, Multiple Dose, Multi-center, Sequential Dose-escalation Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of TB006 in Patients With Mild to Severe Alzheimer's Disease
Brief Title: Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of TB006 in Participants With Alzheimer's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TrueBinding, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: TB006AD2102
Record Dates: First submitted 2021-09-24; First posted 2021-10-12 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Alzheimer's Disease
Keywords: TB006; pharmacokinetics; pharmacodynamics; immunogenicity; mild to severe Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — TB006

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: TB006 (Experimental): Participants will be randomized to 1 of 3 ascending dose groups to receive a total of 5 once-weekly doses of TB006, infused over 1 hour.
  Interventions: Drug: TB006
- Part 1: Placebo (Placebo Comparator): Participants will be randomized to receive 5 once-weekly doses of matching placebo.
  Interventions: Drug: Placebo
- Part 2: TB006 (Experimental): Participants will receive the highest safe and well-tolerated dose identified in Part 1, infused over 1 hour. Randomization will be stratified according to severity at Baseline (mild versus moderate Alzheimer's Disease).
  Interventions: Drug: TB006
- Part 2: Placebo (Placebo Comparator): Participants will be randomized to receive matching placebo. Randomization will be stratified according to severity at Baseline (mild versus moderate Alzheimer's Disease).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TB006 — intravenous infusion
  Arms: Part 1: TB006; Part 2: TB006
Drug: Placebo — intravenous infusion
  Arms: Part 1: Placebo; Part 2: Placebo

SUMMARY:
Part 1 of this study will be conducted to determine the safety, tolerability, and pharmacokinetic (PK) profile of multiple doses of TB006, as well as the maximum tolerated dose of TB006, and to assess the immunogenicity of TB006 (production of anti-TB006 antibody). Part 2 of this study will be conducted to determine the clinical efficacy of TB006 in participants with mild to severe Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Body weight of ≥ 50 kilograms (kg) and body mass index (BMI) between 18 and 35 kg/meters squared (m^2), inclusive
* Mini-Mental State Examination (MMSE) score of 24 or less
* Must be ambulatory
* Clinical diagnosis of Alzheimer's Disease (AD) consistent with the following:

  1. Probable AD, according to National Institute of Neurological and Communicative Disorders and Stroke - Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA)
  2. Meets the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) - Criteria for Major Neurocognitive Disorder (previously dementia)
* Participants or caregiver has the ability to understand the purpose and risks of the study and provide signed and dated informed consent which includes compliance with the requirements and restrictions listed in the inform consent form (ICF) and in this protocol. Participants whose caregiver signs the informed consent must provide their assent.

Exclusion Criteria:

* Any medical or neurological condition other than AD that in the opinion of the investigator could be a contributing cause of the participant's dementia (e.g., medication use, vitamin B12 deficiency, abnormal thyroid function, stroke or other cerebrovascular condition, diffuse Lewy body disease, head trauma)
* History within the past 6 months or evidence of clinically significant psychiatric illness (e.g., major depression, schizophrenia, or bipolar affective disorder)
* Diagnosis of a dementia-related central nervous system (CNS) disease other than AD (e.g., Parkinson's Disease, Huntington's Disease, frontotemporal dementia, multi-infarct dementia, dementia with Lewy bodies, normal pressure hydrocephalus)
* Identification of other known cause of dementia or any other clinically significant contributing co-morbid pathologies at screening magnetic resonance imaging (MRI), in the opinion of the investigator
* Participation in any other drug, biologic, device, or clinical study or treatment with any investigational drug or approved therapy for investigational use within 30 days (or 5 half lives, whichever is longer) prior to screening, and/or participation in any other clinical study involving experimental medications for AD within the 60 days (or 5 half lives, whichever is longer) prior to screening

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: TrueBinding, Inc., Study Director — TrueBinding, Inc.
Locations (14):
- United States (14):
  - Clinical Trial Site, Garden Grove, California
  - Clinical Trial Site, San Diego, California
  - Clinical Trial Site, Delray Beach, Florida
  - Clinical Trial Site, Lady Lake, Florida
  - Clinical Trial Site #1, Maitland, Florida
  - Clinical Trial Site, Maitland, Florida
  - Clinical Trial Site, Miami, Florida
  - Clinical Trial Site, Stuart, Florida
  - Clinical Trial Site, West Palm Beach, Florida
  - Clinical Trial Site, Winter Park, Florida
  - Clinical Trial Site, Decatur, Georgia
  - Clinical Trial Site, Matthews, North Carolina
  - Clinical Trial Site, DeSoto, Texas
  - Clinical Trial Site, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-center study conducted at various centers across United States (US).
Pre-assignment Details: This was a 2-part randomized, double-blind, placebo-controlled, multiple ascending dose (MAD) escalation study that evaluated the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and efficacy of TB006 in participants with Alzheimer's disease (AD).
Groups:
- Part 1: TB006 140 Milligrams (mg) Weekly (qw): Participants were randomized to receive intravenous infusions of TB006 140 mg weekly for over 1 hour.
- Part 1: TB006 420 mg qw: Participants were randomized to receive intravenous infusions of TB006 420 mg weekly for over 1 hour.
- Part 1: TB006 1000 mg qw; Part 2: TB006 1000 mg qw: Participants were randomized to receive intravenous infusions of TB006 1000 mg weekly for over 1 hour.
- Part 1: Placebo; Part 2: Placebo: Participants were randomized to receive intravenous infusions of matching placebo weekly for over 1 hour.
Period: Part 1 (Upto Day 104)
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo | Part 2: TB006 1000 mg qw | Part 2: Placebo
Started | 7 | 6 | 6 | 6 | 0 | 0
Completed | 6 | 6 | 6 | 5 | 0 | 0
Not Completed | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0
Period: Part 2 (Upto Day 104)
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo | Part 2: TB006 1000 mg qw | Part 2: Placebo
Started | 0 | 0 | 0 | 0 | 63 | 66
Completed | 0 | 0 | 0 | 0 | 58 | 64
Not Completed | 0 | 0 | 0 | 0 | 5 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set comprised of all participants randomly assigned to study drug and who took at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo | Part 2: TB006 1000 mg qw | Part 2: Placebo | Total
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 63 | 66 | 154
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.3 (3.25) | 73.0 (10.41) | 71.5 (6.77) | 72.2 (6.74) | 73.5 (9.30) | 71.5 (7.65) | 72.2 (7.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 2 | 5 | 33 | 36 | 86
  Male | 1 | 2 | 4 | 1 | 30 | 30 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 5 | 3 | 27 | 39 | 75
  Not Hispanic or Latino | 7 | 5 | 1 | 3 | 35 | 26 | 77
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 1 | 4 | 6 | 13
  White | 5 | 5 | 6 | 5 | 57 | 60 | 138
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An adverse event is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. An SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, associated with liver injury and impaired liver function or any other situations as per medical or scientific judgement.
Time Frame: Up to Day 104
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 6
Participants
  Any AE | 5 | 4 | 1 | 2
  Any SAE | 1 | 0 | 0 | 0

2. Primary Outcome: Part 1: Change From Baseline in Clinical Chemistry Parameters: Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST) and Creatine Kinase (CK)
Description: Blood samples were collected for analysis of following clinical chemistry parameters including ALT, ALP, AST and CK. Baseline was defined as Day 1. Change from Baseline was obtained by subtracting Baseline value from post-dose visit value.
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: International Units per Liter
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 5
International Units per Liter
  ALT | -1.7 (2.21) | -5.5 (5.32) | -0.7 (10.33) | 5.4 (14.79)
  ALP | -0.6 (9.11) | -4.0 (5.59) | -2.2 (10.05) | 9.0 (15.98)
  AST | -0.1 (2.27) | -3.8 (5.23) | -1.3 (7.61) | 3.2 (13.65)
  CK | 22.0 (39.27) | 0.5 (44.37) | 0.3 (65.56) | -10.4 (14.03)

3. Primary Outcome: Part 1: Change From Baseline in Clinical Chemistry Parameters: Albumin and Protein
Description: Blood samples were collected for analysis of following clinical chemistry parameters including albumin and protein. Baseline was defined as Day 1. Change from Baseline was obtained by subtracting Baseline value from post-dose visit value.
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: grams per deciliter
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 5
grams per deciliter
  Albumin | -0.14 (0.199) | 0.02 (0.098) | -0.03 (0.367) | -0.04 (0.167)
  Protein | -0.20 (0.316) | 0.12 (0.183) | -0.05 (0.589) | -0.08 (0.363)

4. Primary Outcome: Part 1: Change From Baseline in Chemistry Parameters: Calcium, Cholesterol, Creatinine, Direct Bilirubin, Glucose, HDL (High Density Lipoprotein) Cholesterol, LDL (Low Density Lipoprotein) Cholesterol, Total Bilirubin, Triglycerides and Urea Nitrogen
Description: Blood samples were collected for analysis of following clinical chemistry parameters including Calcium, Cholesterol, Creatinine, Direct Bilirubin, Glucose, HDL Cholesterol, LDL Cholesterol, Total Bilirubin, Triglycerides and Urea Nitrogen. Baseline was defined as Day 1. Change from Baseline was obtained by subtracting Baseline value from post-dose visit value.
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 5
milligrams per deciliter
  Calcium | -0.13 (0.373) | 0.17 (0.280) | -0.02 (0.360) | -0.18 (0.356)
  Cholesterol | -15.4 (21.62) | -2.7 (10.35) | 6.2 (74.37) | -13.4 (47.79)
  Creatinine | 0.047 (0.081) | 0.153 (0.377) | 0.108 (0.143) | -0.040 (0.142)
  Direct Bilirubin | -0.007 (0.032) | -0.003 (0.033) | 0.000 (0.020) | -0.022 (0.030)
  Glucose | 34.3 (55.23) | -15.0 (18.51) | 21.3 (45.45) | 8.2 (49.94)
  HDL Cholesterol | -3.6 (5.19) | -3.0 (4.65) | 0.2 (13.98) | 4.0 (17.13)
  LDL Cholesterol | -9.0 (9.04) | -1.8 (9.33) | -3.5 (64.62) | -14.8 (46.23)
  Total Bilirubin | -0.036 (0.093) | -0.005 (0.227) | 0.032 (0.132) | -0.134 (0.225)
  Triglycerides | -23.3 (69.65) | 12.2 (17.72) | 18.7 (104.95) | -23.8 (39.06)
  Urea Nitrogen | -0.40 (2.171) | 6.95 (8.277) | 2.43 (3.449) | 1.30 (4.266)

5. Primary Outcome: Part 1: Change From Baseline in Clinical Chemistry Parameter: Hemoglobin A1C
Description: Blood samples were collected for analysis of following clinical chemistry parameters including Hemoglobin A1C. Baseline was defined as Day 1. Change from Baseline was obtained by subtracting Baseline value from post-dose visit value.
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 5
percentage of glycosylated hemoglobin | 0.06 (0.162) | -0.02 (0.567) | -0.33 (0.625) | -0.14 (1.011)

6. Primary Outcome: Part 1: Change From Baseline in Clinical Chemistry Parameters: Potassium and Sodium
Description: Blood samples were collected for analysis of following clinical chemistry parameters including Potassium and Sodium. Baseline was defined as Day 1. Change from Baseline was obtained by subtracting Baseline value from post-dose visit value.
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 5
Millimoles per liter
  Potassium | 0.10 (0.476) | -0.15 (0.288) | 0.07 (0.378) | 0.02 (0.259)
  Sodium | -1.0 (2.24) | 0.8 (1.72) | -1.2 (2.56) | -1.2 (2.39)

7. Primary Outcome: Part 1: Change From Baseline in Clinical Chemistry Parameter: Thyrotropin
Description: Blood samples were collected for analysis of following clinical chemistry parameters including Thyrotropin. Baseline was defined as Day 1. Change from Baseline was obtained by subtracting Baseline value from post-dose visit value.
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: micro-international units per milliliter
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 5
micro-international units per milliliter | 1.209 (3.114) | -0.343 (0.298) | -0.370 (1.312) | -0.246 (0.372)

8. Primary Outcome: Part 1: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils and Platelets
Description: Blood samples were collected for analysis of following hematology parameters including Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils and Platelets. Baseline was defined as Day 1. Change from Baseline was obtained by subtracting Baseline value from post-dose visit value.
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: 10^3 cells per microliter
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 5
10^3 cells per microliter
  Basophils | -0.023 (0.015) | -0.005 (0.019) | 0.005 (0.028) | 0.006 (0.013)
  Eosinophils | 0.014 (0.138) | 0.003 (0.068) | 0.038 (0.089) | 0.030 (0.173)
  Leukocytes | -0.76 (0.650) | 0.00 (1.292) | 0.40 (1.563) | -0.28 (1.092)
  Lymphocytes | -0.264 (0.188) | -0.025 (0.241) | -0.037 (1.265) | -0.036 (0.250)
  Monocytes | -0.094 (0.118) | -0.017 (0.114) | 0.032 (0.108) | 0.028 (0.062)
  Neutrophils | -0.396 (0.719) | 0.078 (1.171) | 0.368 (0.641) | -0.318 (1.145)
  Platelets: number analyzed (Participants) | 7 | 6 | 5 | 4
  Platelets | -9.1 (37.53) | 5.0 (37.25) | -9.6 (89.83) | -4.5 (50.16)

9. Primary Outcome: Part 1: Change From Baseline in Hematology Parameter: Erythrocyte. Mean Corpuscular Hemoglobin (Ery. MCH)
Description: Blood samples were collected for analysis of following hematology parameter: Ery. MCH. Baseline was defined as Day 1. Change from Baseline was obtained by subtracting Baseline value from post-dose visit value.
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: picograms
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 5
picograms | -0.40 (1.134) | -0.05 (0.579) | 1.02 (3.511) | -0.34 (0.631)

10. Primary Outcome: Part 1: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected for analysis of following hematology parameter: Hematocrit. Baseline was defined as Day 1. Change from Baseline was obtained by subtracting Baseline value from post-dose visit value.
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 5
Percentage | 0.69 (2.563) | 1.18 (2.105) | 1.18 (7.919) | 0.32 (2.493)

11. Primary Outcome: Part 1: Change From Baseline in Hematology Parameter: Erythrocytes and Reticulocytes
Description: Blood samples were collected for analysis of following hematology parameter: Erythrocytes and Reticulocytes. Baseline was defined as Day 1. Change from Baseline was obtained by subtracting Baseline value from post-dose visit value.
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: 10^6 cells per microliter
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 5
10^6 cells per microliter
  Erythrocytes | 0.039 (0.401) | 0.012 (0.219) | -0.108 (0.625) | 0.024 (0.211)
  Reticulocytes | -0.011 (0.017) | -0.005 (0.004) | -0.008 (0.008) | -0.005 (0.009)

12. Primary Outcome: Part 1: Change From Baseline in Hematology Parameter: Erythrocyte. Mean Corpuscular Volume (Ery. MCV)
Description: Blood samples were collected for analysis of following hematology parameter: Ery. MCV. Baseline was defined as Day 1. Change from Baseline was obtained by subtracting Baseline value from post-dose visit value.
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: femtoliters
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 5
femtoliters | 0.80 (1.926) | 2.45 (1.343) | 5.42 (5.724) | 0.20 (2.699)

13. Primary Outcome: Part 1: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were collected for analysis of following hematology parameter: Baseline was defined as Day 1. Change from Baseline was obtained by subtracting Baseline value from post-dose visit value.
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: grams per deciliter
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 5
grams per deciliter | -0.06 (0.779) | 0.00 (0.465) | 0.08 (3.260) | -0.10 (0.877)

14. Primary Outcome: Part 1: Change From Baseline in Urine Potential of Hydrogen (pH)
Description: Urine samples were collected for analysis of Urine pH. Baseline was defined as Day 1. Change from Baseline was obtained by subtracting Baseline value from post-dose visit value.
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: potential of Hydrogen
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo
Number analyzed (Participants) | 7 | 5 | 6 | 5
potential of Hydrogen | -0.36 (1.215) | 0.40 (1.294) | -0.50 (1.612) | -0.80 (0.975)

15. Primary Outcome: Part 1: Change From Baseline in Urine Specific Gravity
Description: Urine samples were collected for analysis of Urine specific gravity. Baseline was defined as Day 1. Change from Baseline was obtained by subtracting Baseline value from post-dose visit value.
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo
Number analyzed (Participants) | 7 | 5 | 6 | 5
Ratio | 0.003 (0.008) | 0.003 (0.006) | 0.004 (0.011) | 0.007 (0.010)

16. Primary Outcome: Part 1: Change From Baseline in Urobilinogen
Description: Urine samples were collected for analysis of Urobilinogen. Baseline was defined as Day 1. Change from Baseline was obtained by subtracting Baseline value from post-dose visit value.
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo
Number analyzed (Participants) | 7 | 5 | 6 | 5
milligrams per deciliter | 0.00 (0.462) | -0.16 (0.358) | -0.13 (0.602) | 0.00 (0.000)

17. Primary Outcome: Part 1: Change From Baseline in Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: Vital signs including DBP and SBP was measured by at least 5 minutes of rest with the participant in a quiet setting without distractions (eg, television, cell phones). Blood pressure measurements were taken with the participant in the sitting position. Baseline was defined as the last available value prior to the participant receiving the first study drug infusion on Day 1. Change from Baseline was obtained by subtracting the Baseline value from post-dose visit value.
Time Frame: Baseline and Up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 5
Millimeters of mercury
  DBP | -2.1 (12.06) | -2.3 (10.37) | -1.0 (3.03) | -7.2 (9.09)
  SBP | -10.4 (13.39) | 3.5 (9.61) | -6.2 (13.17) | 2.2 (17.74)

18. Primary Outcome: Part 1: Change From Baseline in Respiratory Rate
Description: Vital signs including respiratory rate was measured by at least 5 minutes of rest with the participant in a quiet setting without distractions (eg, television, cell phones). Baseline was defined as the last available value prior to the participant receiving the first study drug infusion on Day 1. Change from Baseline was obtained by subtracting the Baseline value from post-dose visit value.
Time Frame: Baseline and Up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 5
breaths per minute | 0.0 (0.00) | -0.7 (2.16) | 0.3 (1.03) | -0.2 (1.30)

19. Primary Outcome: Part 1: Change From Baseline in Temperature
Description: Vital signs including temperature was measured by at least 5 minutes of rest with the participant in a quiet setting without distractions (eg, television, cell phones). Baseline was defined as the last available value prior to the participant receiving the first study drug infusion on Day 1. Change from Baseline was obtained by subtracting the Baseline value from post-dose visit value.
Time Frame: Baseline and Up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 5
degrees Celsius | 0.26 (0.351) | -0.37 (0.350) | -0.03 (0.833) | -0.22 (0.130)

20. Primary Outcome: Part 1: Change From Baseline in Heart Rate
Description: Vital signs including heart rate was measured by at least 5 minutes of rest with the participant in a quiet setting without distractions (eg, television, cell phones). Baseline was defined as the last available value prior to the participant receiving the first study drug infusion on Day 1. Change from Baseline was obtained by subtracting the Baseline value from post-dose visit value.
Time Frame: Baseline and Up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 5
Beats per minute | -2.0 (8.00) | 3.3 (3.72) | 4.0 (5.73) | -4.2 (9.50)

21. Primary Outcome: Part 1: Change From Baseline in Electrocardiogram (ECG) Mean Heart Rate
Description: 12-lead ECG measurements was obtained using an ECG machine that automatically calculates the heart rate. Baseline was defined as the last available value prior to the participant receiving the first study drug infusion on Day 1. Change from Baseline was obtained by subtracting the Baseline value from post-dose visit value value.
Time Frame: Baseline and Up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 5
Beats per minute | -4.8 (5.78) | -0.9 (4.00) | 3.0 (3.82) | -3.4 (4.87)

22. Primary Outcome: Part 1: Change From Baseline in ECG Parameters
Description: 12-lead ECG measurements was obtained using an ECG machine that automatically calculates the PR interval, QRS duration, QT interval and QT Corrected using Bazett's formula (QTcB). Baseline was defined as the last available value prior to the participant receiving the first study drug infusion on Day 1. Change from Baseline was obtained by subtracting the Baseline value from post-dose visit value.
Time Frame: Baseline and Up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 5
milliseconds
  PR Interval | 4.8 (10.07) | 0.7 (5.90) | -11.0 (14.74) | 14.9 (5.16)
  QRS Duration | 0.3 (3.07) | 1.1 (5.27) | 1.0 (7.16) | -4.1 (13.50)
  QT Interval | 21.9 (12.72) | -2.9 (10.48) | 0.3 (9.36) | -5.0 (11.47)
  QTcB Interval | 8.1 (11.37) | -6.6 (12.98) | 9.9 (11.50) | -15.2 (4.15)

23. Primary Outcome: Part 1: Number of Participants With Suicidal Ideation or Suicidal Behavior as Measured Using Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is an interview-based instrument to systematically assess suicidal ideation and suicidal behavior. Number of participants that have an affirmative response to the 5 items for suicidal ideation (1. Wish to be dead, 2. Non-specific active suicidal thoughts, 3. Active suicidal ideation with any methods without intent to act, 4. Active suicidal ideation with some intent to act, without specific plan, 5. Active suicidal ideation with specific plan and intent) and/or to the 5 items for suicidal behavior (1. Preparatory acts or behavior, 2. Aborted attempt, 3. Interrupted attempt, 4. Actual attempt, 5. Completed suicide) were reported. The total score ranges from 0 (no ideation present) to 5 (active suicidal ideation with specific plan and intent); higher scores indicate worse symptoms.
Time Frame: Up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 5
Participants
  Wish to be dead | 0 | 0 | 0 | 0
  Non-specific active suicidal thoughts | 0 | 0 | 0 | 0
  Active suicidal ideation without any methods without intent to act | 0 | 0 | 0 | 0
  Active suicidal ideation with some intent to act, without specific plan | 0 | 0 | 0 | 0
  Active suicidal ideation with specific plan and intent | 0 | 0 | 0 | 0
  Any suicidal behavior | 0 | 0 | 0 | 0
  Actual attempt | 0 | 0 | 0 | 0
  Interrupted attempt | 0 | 0 | 0 | 0
  Aborted attempt | 0 | 0 | 0 | 0
  Preparatory acts or behavior | 0 | 0 | 0 | 0
  Most recent attempt | 0 | 0 | 0 | 0
  First attempt | 0 | 0 | 0 | 0
  Lethal attempt | 0 | 0 | 0 | 0

24. Primary Outcome: Part 1: Number of Participants With Clinically Significant Physical Examination Findings
Description: A complete physical examination included, at a minimum, assessment of the Cardiovascular, Respiratory, Gastrointestinal and Neurological systems. This analysis was planned but data was not captured in the database. Abnormal changes were captured as adverse events if they were clinically significant.
Time Frame: Up to Day 104
Population: Full analysis set comprised of all participants who are randomly assigned to study drug. This analysis was planned but data was not captured in the database.
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

25. Primary Outcome: Part 1: Number of Participants With Clinically Significant Neurological Examination Findings
Description: The neurological examination assessed mental status, motor and sensory skills, hearing and speech, vision, coordination, and balance. This analysis was planned but data was not captured in the database. Abnormal changes were captured as adverse events if they were clinically significant.
Time Frame: Up to Day 104
Population: Full Analysis Set. This analysis was planned but data was not captured in the database.
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

26. Primary Outcome: Part 1: Dose Normalized Area Under the Concentration Time Curve Over a Dosing Interval (AUCtau) of TB006
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of TB006. PK parameters were analyzed using standard non-compartmental analysis. AUCtau normalized to the actual administered dose is presented. The AUCtau was divided by the actual dose strength to get the normalized area under the concentration-time curve.
Time Frame: Day 1 and Day 29
Population: Pharmacokinetic Analysis Set comprises of all participants who received at least 1 dose of TB006 and have at least 1 post-dose blood sample with measurable TB006 concentrations. Only those participants with data available at specified timepoints has been presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*micrograms/milliliter/milligram
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw
Number analyzed (Participants) | 7 | 6 | 5
hours*micrograms/milliliter/milligram
  Day 1: number analyzed (Participants) | 6 | 5 | 2
  Day 1 | 39.81 (23.17) | 29.87 (38.15) | 11.93 (100.21)
  Day 29 | 125.92 (18.01) | 117.75 (24.52) | 82.95 (18.18)

27. Primary Outcome: Part 1: Time at Which Maximum Plasma Concentration Occurs (Tmax) of TB006
Description: Blood samples were collected at indicated time points for PK analysis of TB006. PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: At Days 1, 8 and 29
Population: Pharmacokinetic Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw
Number analyzed (Participants) | 7 | 6 | 6
hours
  Day 1 | 1.12 [1.0 to 7.0] | 2.01 [1.1 to 5.0] | 2.00 [1.0 to 5.0]
  Day 8 | 1.23 [1.0 to 2.0] | 1.60 [1.2 to 5.0] | 2.50 [1.1 to 5.0]
  Day 29: number analyzed (Participants) | 7 | 6 | 5
  Day 29 | 2.03 [1.1 to 5.1] | 2.18 [1.1 to 7.0] | 2.00 [1.0 to 7.0]

28. Primary Outcome: Part 1: Dose Normalized Maximum Observed Plasma Concentration (Cmax) of TB006
Description: Blood samples were collected at indicated time points for PK analysis of TB006. PK parameters were analyzed using standard non-compartmental analysis. Cmax normalized to the actual administered dose is presented. The Cmax was divided by the actual dose strength to get the normalized maximum observed plasma concentration.
Time Frame: At Days 1, 8 and 29
Population: Pharmacokinetic Analysis Set. Only those participants with data available at specified timepoints has been presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter/milligram
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw
Number analyzed (Participants) | 7 | 6 | 6
micrograms/milliliter/milligram
  Day 1 | 0.36 (25.72) | 0.29 (36.97) | 0.07 (105.32)
  Day 8 | 0.58 (27.57) | 0.49 (26.77) | 0.30 (30.27)
  Day 29: number analyzed (Participants) | 7 | 6 | 5
  Day 29 | 0.95 (18.15) | 0.85 (22.89) | 0.61 (13.40)

29. Primary Outcome: Part 1: Concentration at the End of a Dosing Interval (Ctrough) of TB006
Description: as for outcome 27
Time Frame: Day 8 and Day 29
Population: Pharmacokinetic Analysis Set. Only those participants with data available at specified timepoints has been presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw
Number analyzed (Participants) | 7 | 6 | 5
micrograms per milliliter
  Day 8: number analyzed (Participants) | 7 | 5 | 3
  Day 8 | 25.77 (21.23) | 71.44 (20.75) | 68.62 (70.91)
  Day 29 | 76.69 (19.62) | 204.77 (20.46) | 348.20 (22.34)

30. Primary Outcome: Part 1: Terminal Elimination Phase Half-life (t1/2) of TB006
Description: as for outcome 27
Time Frame: At Day 29
Population: Pharmacokinetic Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw
Number analyzed (Participants) | 7 | 6 | 4
hours | 711.49 (19.87) | 757.59 (22.80) | 739.50 (14.90)

31. Primary Outcome: Part 1: Total Clearance (CL) of TB006
Description: as for outcome 27
Time Frame: At Day 29
Population: Pharmacokinetic Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliters per hour
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw
Number analyzed (Participants) | 7 | 6 | 5
milliliters per hour | 7.94 (17.06) | 8.49 (19.27) | 12.06 (19.68)

32. Primary Outcome: Part 1: Volume of Distribution (Vd) of TB006
Description: as for outcome 27
Time Frame: At Day 29
Population: Pharmacokinetic Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliters
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw
Number analyzed (Participants) | 7 | 6 | 4
milliliters | 8151.47 (21.38) | 9282.51 (28.97) | 13617.70 (30.63)

33. Primary Outcome: Part 1: Number of Participants With Anti-TB006 Antibodies (Immunogenicity of TB006)
Description: Plasma samples were collected at indicated time points for the determination of anti-TB006 antibodies. Plasma samples were screened for antibodies binding to TB006 and the titer of confirmed positive samples has been reported.
Time Frame: Day 1 (Predose), Day 8 (Predose), Day 36 and Day 104
Population: Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo
Number analyzed (Participants) | 7 | 6 | 6 | 6
Participants
  Day 1 (Predose) | 0 | 0 | 0 | 0
  Day 8 (Predose) | 0 | 0 | 0 | 0
  Day 36 | 0 | 0 | 0 | 0
  Day 104 | 1 | 0 | 0 | 0

34. Primary Outcome: Part 2: Change From Baseline Through Day 104 on the Clinical Dementia Rating Scale - Sum of Boxes Total Score
Description: The Clinical Dementia Rating was obtained through semi-structured interviews of participants and informants, and cognitive functioning was rated in six domains of functioning: memory, orientation, judgement and problem solving, community affairs, home and hobbies, and personal care. Each domain was rated on a five-point scale of functioning as follows: 0: no impairment; 0.5: questionable impairment; 1: mild impairment; 2: moderate impairment; and 3: severe impairment. The Clinical Dementia Rating Scale - Sum of Boxes was based on summing each of the domain box scores with total scores ranging from 0-18, where lower total scores represent better outcomes, and higher total scores represent worse outcomes. Baseline was defined as the last available value prior to the subject receiving the first study drug infusion on Day 1. Change from Baseline value was obtained by subtracting Baseline value from post-dose visit value.
Time Frame: Baseline through Day 104
Population: Efficacy Analysis Set comprised of all participants who received assigned dose of TB006 in Part 2 and the participants enrolled at the same TB006 dose level in Part 1, as well as all placebo participants were included and had at least one post-dose evaluable Pharmacodynamic assessment across participant.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 67 | 72
Scores on a scale | 0.01 (0.147) | 0.35 (0.142)
Statistical Analysis 1: Comparison: Part 2: TB006 1000 mg qw vs Part 2: Placebo; Test type: Other; p = 0.0838, Mixed Models Analysis; Least square mean difference = -0.35, 95% CI 2-sided [-0.741 to 0.047]

35. Secondary Outcome: Part 2: Change From Baseline Through Day 36 on the Clinical Dementia Rating Scale - Sum of Boxes Total Score
Description: as for outcome 34
Time Frame: Baseline through Day 36
Population: Efficacy Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 67 | 72
Scores on a scale | -0.16 (0.162) | 0.23 (0.157)

36. Secondary Outcome: Part 2: Percentage of Responders on the Clinical Dementia Rating Scale - Sum of Boxes
Description: The Clinical Dementia Rating is obtained through semi-structured interviews of participants and informants, and cognitive functioning is rated in six domains of functioning: memory, orientation, judgement and problem solving, community affairs, home and hobbies, and personal care. Each domain is rated on a five-point scale of functioning as follows: 0, no impairment; 0.5, questionable impairment; 1, mild impairment; 2, moderate impairment; and 3, severe impairment. The Clinical Dementia Rating Scale - Sum of Boxes is based on summing each of the domain box scores with total scores ranging from 0-18, where lower total scores represent better outcomes, and higher total scores represent worse outcomes. A responder was defined as a participant with at least 1 point improvement from Baseline on the Sum of Boxes score. Percentage of responders on the Clinical Dementia Rating Scale - Sum of Boxes has been presented.
Time Frame: At Days 36 and 104
Population: Efficacy Analysis Set.
Measure: Number; unit: Percentage of responders
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 67 | 72
Percentage of responders
  Day 36 | 25.4 | 9.7
  Day 104 | 22.4 | 15.3

37. Secondary Outcome: Part 2: Change From Baseline on Mini-Mental State Examination (MMSE) Score
Description: The MMSE was used to measure cognitive impairment. The MMSE can evaluate overall cognitive function, and is widely used for the assessment of cognitive impairment in dementia participants. The questionnaire consists of 11 items, and each item aims to evaluate different cognitive domains such as orientation, memory, attention, and construction. The score ranged from 0 to 30, with a higher score indicating better function. A positive change score indicated improvement from Baseline. Baseline was defined as Day 1. Change from Baseline was obtained by subtracting Baseline value from post-dose visit value.
Time Frame: Baseline and at Days 36 and 104
Population: Efficacy Analysis Set. Only those participants with data available at specified timepoints has been presented.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 66 | 70
Scores on a scale
  Day 36 | 1.2 (2.59) | 0.2 (2.52)
  Day 104: number analyzed (Participants) | 63 | 69
  Day 104 | 1.0 (3.10) | 0.6 (2.97)

38. Secondary Outcome: Part 2: Change From Baseline on the Neuropsychiatric Inventory (NPI) Score
Description: The NPI was a questionnaire that quantified psychiatric symptoms and behavioral disorders in dementia. A total of 12 items (the original NPI-10 consisting of 10 behavioral domains: delusions, hallucinations, agitation/aggression, dysphoria, anxiety, euphoria, apathy, disinhibition, irritability/lability, and aberrant motor behavior, The NPI total score was calculated by adding the scores of the domains (each domain scores ranges from 0 to 12). The NPI total score ranges from 0 to 120 with higher scores indicating greater behavioral impairment. Baseline was defined as Day 1. Change from Baseline was obtained by subtracting Baseline value from post-dose visit value.
Time Frame: Baseline and at Days 36 and 104
Population: Efficacy Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 66 | 69
Scores on a scale
  Day 36 | -2.5 (8.10) | -0.8 (9.12)
  Day 104: number analyzed (Participants) | 63 | 69
  Day 104 | -3.5 (11.47) | -1.1 (6.79)

39. Secondary Outcome: Part 2: Number of Participants With AEs and SAEs
Description: as for outcome 1
Time Frame: Up to Day 104
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 63 | 66
Participants
  Any AE | 28 | 17
  Any SAE | 4 | 1

40. Secondary Outcome: Part 2: Change From Baseline in Clinical Chemistry Parameters: ALT, ALP, AST and CK
Description: as for outcome 2
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: International Units per Liter
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 58 | 64
International Units per Liter
  ALT | -0.5 (12.88) | -0.4 (5.40)
  ALP | 1.0 (12.01) | 0.0 (11.92)
  AST | -0.4 (10.44) | -0.5 (3.58)
  CK | -14.3 (77.24) | 6.3 (52.07)

41. Secondary Outcome: Part 2: Change From Baseline in Clinical Chemistry Parameters: Albumin and Protein
Description: as for outcome 3
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: grams per deciliter
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 58 | 64
grams per deciliter
  Albumin | -0.10 (0.300) | -0.01 (0.251)
  Protein | -0.10 (0.470) | 0.00 (0.404)

42. Secondary Outcome: Part 2: Change From Baseline in Chemistry Parameters: Calcium, Cholesterol, Creatinine, Direct Bilirubin, Glucose, HDL Cholesterol, LDL Cholesterol, Total Bilirubin, Triglycerides and Urea Nitrogen
Description: as for outcome 4
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 58 | 64
milligrams per deciliter
  Calcium | -0.09 (0.437) | -0.11 (0.432)
  Cholesterol | -5.8 (32.30) | 0.3 (28.17)
  Creatinine | 0.014 (0.098) | -0.017 (0.124)
  Direct Bilirubin | 0.005 (0.037) | -0.006 (0.030)
  Glucose | -5.6 (26.98) | -6.3 (27.92)
  HDL Cholesterol | -2.4 (8.49) | -0.3 (8.26)
  LDL Cholesterol | -7.5 (24.64) | -4.6 (23.63)
  Total Bilirubin | 0.023 (0.157) | -0.014 (0.128)
  Triglycerides | -9.2 (73.95) | -0.4 (46.29)
  Urea Nitrogen | 0.41 (3.817) | -1.03 (4.777)

43. Secondary Outcome: Part 2: Change From Baseline in Clinical Chemistry Parameter: Hemoglobin A1C
Description: Blood samples were collected for analysis of following clinical chemistry parameter including Hemoglobin A1C. Baseline was defined as Day 1. Change from Baseline was obtained by subtracting Baseline value from post-dose visit value.
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 54 | 63
percentage of glycosylated hemoglobin | -0.06 (0.638) | 0.07 (0.555)

44. Secondary Outcome: Part 2: Change From Baseline in Clinical Chemistry Parameters: Potassium and Sodium
Description: as for outcome 6
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 58 | 64
Millimoles per liter
  Potassium | -0.14 (0.469) | -0.13 (0.521)
  Sodium | -0.7 (2.11) | -0.7 (3.05)

45. Secondary Outcome: Part 2: Change From Baseline in Clinical Chemistry Parameter: Thyrotropin
Description: Blood samples were collected for analysis of following clinical chemistry parameter including Thyrotropin. Baseline was defined as Day 1. Change from Baseline was obtained by subtracting Baseline value from post-dose visit value.
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: micro-international units per milliliter
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 58 | 64
micro-international units per milliliter | -0.118 (0.619) | 0.134 (1.000)

46. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Leukocytes, Lymphocytes, Monocytes, Neutrophils and Platelets
Description: as for outcome 8
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: 10^3 cells per microliter
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 58 | 63
10^3 cells per microliter
  Basophils | -0.004 (0.027) | -0.002 (0.022)
  Eosinophils | -0.008 (0.113) | -0.040 (0.130)
  Leukocytes | -0.26 (1.383) | -0.02 (1.244)
  Lymphocytes | -0.118 (0.392) | -0.053 (0.411)
  Monocytes | -0.021 (0.109) | 0.003 (0.107)
  Neutrophils | -0.109 (1.295) | 0.067 (1.206)
  Platelets: number analyzed (Participants) | 57 | 61
  Platelets | -1.9 (32.08) | -12.1 (46.27)

47. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Ery. MCH
Description: as for outcome 9
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: picograms
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 58 | 63
picograms | 0.19 (0.775) | 0.51 (1.045)

48. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Ery. MCV
Description: as for outcome 12
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: femtoliters
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 58 | 63
femtoliters | 1.54 (2.743) | 2.04 (3.412)

49. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Erythrocytes and Reticulocytes
Description: as for outcome 11
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: 10^6 cells per microliter
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 58 | 63
10^6 cells per microliter
  Erythrocytes | -0.028 (0.269) | 0.024 (0.228)
  Reticulocytes | 0.001 (0.012) | -0.003 (0.012)

50. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Hematocrit
Description: as for outcome 10
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 58 | 63
Percentage | 0.41 (2.735) | 1.11 (2.403)

51. Secondary Outcome: Part 2: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were collected for analysis of following hematology parameter: Hemoglobin. Baseline was defined as Day 1. Change from Baseline was obtained by subtracting Baseline value from post-dose visit value.
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: grams per deciliter
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 58 | 63
grams per deciliter | 0.00 (0.766) | 0.29 (0.827)

52. Secondary Outcome: Part 2: Change From Baseline in Urine pH
Description: as for outcome 14
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: potential of Hydrogen
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 57 | 61
potential of Hydrogen | -0.13 (0.788) | 0.18 (0.791)

53. Secondary Outcome: Part 2: Change From Baseline in Urine Specific Gravity
Description: as for outcome 15
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 57 | 61
Ratio | 0.002 (0.010) | 0.001 (0.008)

54. Secondary Outcome: Part 2: Change From Baseline in Urobilinogen
Description: as for outcome 16
Time Frame: Baseline and up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 57 | 61
milligrams per deciliter | 0.07 (0.313) | 0.05 (0.354)

55. Secondary Outcome: Part 2: Change From Baseline in DBP and SBP
Description: as for outcome 17
Time Frame: Baseline and Up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 58 | 64
Millimeters of mercury
  DBP | 0.8 (6.42) | 0.7 (9.48)
  SBP | 1.4 (15.02) | 0.0 (15.57)

56. Secondary Outcome: Part 2: Change From Baseline in Respiratory Rate
Description: Vital signs including respiratory rate was measured by at least 5 minutes of rest with the participant in a quiet setting without distractions (eg, television, cell phones). Blood pressure measurements were taken with the participant in the sitting position. Baseline was defined as the last available value prior to the participant receiving the first study drug infusion on Day 1. Change from Baseline was obtained by subtracting the Baseline value from post-dose visit value.
Time Frame: Baseline and Up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 58 | 64
breaths per minute | 0.1 (0.97) | 0.2 (0.97)

57. Secondary Outcome: Part 2: Change From Baseline in Temperature
Description: Vital signs including temperature was measured by at least 5 minutes of rest with the participant in a quiet setting without distractions (eg, television, cell phones). Blood pressure measurements were taken with the participant in the sitting position. Baseline was defined as the last available value prior to the participant receiving the first study drug infusion on Day 1. Change from Baseline was obtained by subtracting the Baseline value from post-dose visit value.
Time Frame: Baseline and Up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 58 | 64
degrees Celsius | 0.01 (0.489) | -0.03 (0.461)

58. Secondary Outcome: Part 2: Change From Baseline in Heart Rate
Description: Vital signs including heart rate was measured by at least 5 minutes of rest with the participant in a quiet setting without distractions (eg, television, cell phones). Blood pressure measurements were taken with the participant in the sitting position. Baseline was defined as the last available value prior to the participant receiving the first study drug infusion on Day 1. Change from Baseline was obtained by subtracting the Baseline value from post-dose visit value.
Time Frame: Baseline and Up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 58 | 64
Beats per minute | -4.2 (8.59) | -2.1 (7.86)

59. Secondary Outcome: Part 2: Change From Baseline in ECG Parameters
Description: 12-lead ECG measurements was obtained using an ECG machine that automatically calculates the PR interval, QRS duration, QT interval and QTcB. Baseline was defined as the last available value prior to the participant receiving the first study drug infusion on Day 1. Change from Baseline was obtained by subtracting the Baseline value from post-dose visit value.
Time Frame: Baseline and Up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 58 | 63
milliseconds
  PR Interval: number analyzed (Participants) | 57 | 63
  PR Interval | -1.6 (13.17) | 2.1 (18.32)
  QRS Duration | -2.2 (13.31) | -1.4 (7.71)
  QT Interval | 4.2 (26.29) | 3.9 (20.28)
  QTcB Interval | -2.0 (18.01) | -1.7 (15.99)

60. Secondary Outcome: Part 2: Change From Baseline in ECG Mean Heart Rate
Description: 12-lead ECG measurements was obtained using an ECG machine that automatically calculates the heart rate. Baseline was defined as the last available value prior to the participant receiving the first study drug infusion on Day 1. Change from Baseline was obtained by subtracting the Baseline value from post-dose visit value.
Time Frame: Baseline and Up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 58 | 63
Beats per minute | -1.8 (8.87) | -1.3 (7.40)

61. Secondary Outcome: Part 2: Number of Participants With Suicidal Ideation or Suicidal Behavior as Measured Using C-SSRS
Description: as for outcome 23
Time Frame: Up to Day 104
Population: Safety Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 58 | 64
Participants
  Wish to be dead | 0 | 0
  Non-specific active suicidal thoughts | 0 | 0
  Active suicidal ideation without any methods without intent to act | 0 | 0
  Active suicidal ideation with some intent to act, without specific plan | 0 | 0
  Active suicidal ideation with specific plan and intent | 0 | 0
  Any suicidal behavior | 0 | 0
  Actual attempt | 0 | 0
  Interrupted attempt | 0 | 0
  Aborted attempt | 0 | 0
  Preparatory acts or behavior | 0 | 0
  Most recent attempt | 0 | 0
  First attempt | 0 | 0
  Lethal attempt | 0 | 0

62. Secondary Outcome: Part 2: Number of Participants With Clinically Significant Physical Examination Findings
Description: as for outcome 24
Time Frame: Up to Day 104
Population: Full Analysis Set. This analysis was planned but data was not captured in the database.
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 0 | 0

63. Secondary Outcome: Part 2: Number of Participants With Clinically Significant Neurological Examination Findings
Description: as for outcome 25
Time Frame: Up to Day 104
Population: Full Analysis Set. This analysis was planned but data was not captured in the database.
Arm/Group | Part 2: TB006 1000 mg qw | Part 2: Placebo
Number analyzed (Participants) | 0 | 0

64. Secondary Outcome: Part 2: Ctrough of TB006
Description: as for outcome 27
Time Frame: Day 29
Population: Pharmacokinetic Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter
Arm/Group | Part 2: TB006 1000 mg qw
Number analyzed (Participants) | 59
micrograms per milliliter | 395.82 (35.88)

65. Secondary Outcome: Part 2: t1/2 of TB006
Description: as for outcome 27
Time Frame: Day 29
Population: Pharmacokinetic Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 2: TB006 1000 mg qw
Number analyzed (Participants) | 48
hours | 756.78 (22.05)

66. Secondary Outcome: Part 2: Cmax of TB006
Description: as for outcome 27
Time Frame: Day 1 and Day 29
Population: Pharmacokinetic Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 2: TB006 1000 mg qw
Number analyzed (Participants) | 58
Micrograms per milliliter
  Day 1 | 339.17 (23.82)
  Day 29: number analyzed (Participants) | 56
  Day 29 | 731.55 (25.13)

ADVERSE EVENTS:
Time Frame: Up to Day 104
Description: Serious adverse events and non-Serious adverse events were collected in Safety Analysis Set and comprised of all participants randomly assigned to study drug and who took at least 1 dose of study drug.
Arm/Group | Part 1: TB006 140 Milligrams (mg) Weekly (qw) | Part 1: TB006 420 mg qw | Part 1: TB006 1000 mg qw | Part 1: Placebo | Part 2: TB006 1000 mg qw | Part 2: Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/6 | 0/6 | 1/63 | 0/66
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/6 | 0/6 | 0/6 | 4/63 | 1/66
Other Adverse Events (participants affected / at risk) | 5/7 | 4/6 | 1/6 | 2/6 | 28/63 | 17/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: TB006 140 Milligrams (mg) Weekly (qw) (N=7) | Part 1: TB006 420 mg qw (N=6) | Part 1: TB006 1000 mg qw (N=6) | Part 1: Placebo (N=6) | Part 2: TB006 1000 mg qw (N=63) | Part 2: Placebo (N=66)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: TB006 140 Milligrams (mg) Weekly (qw) (N=7) | Part 1: TB006 420 mg qw (N=6) | Part 1: TB006 1000 mg qw (N=6) | Part 1: Placebo (N=6) | Part 2: TB006 1000 mg qw (N=63) | Part 2: Placebo (N=66)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Thyroid function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine analysis abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Claustrophobia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/98/NCT05074498/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-14): https://cdn.clinicaltrials.gov/large-docs/98/NCT05074498/SAP_002.pdf